CLINICAL TRIAL: NCT04101266
Title: Comparison of the Effects Combined Suprascapular and Infraclavicular Nerve Blocks to Interscalene Nerve Block Applied Arthtroscopic Shoulder Surgery
Brief Title: Pain Management in Arthtroscopic Shoulder Surgery
Acronym: PMSS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Diskapi Yildirim Beyazit Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Tugba Arslan, Principle Investigator, Diskapi Yildirim Beyazit Education and Research Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 59/13
Record Dates: First submitted 2019-09-17; First posted 2019-09-24 (Actual); Last update posted 2021-06-10 (Actual); Status verified 2021-06

CONDITIONS: Arthroscopic Shoulder Surgery

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interscalene nerve block (Active Comparator): preoperative interscalene nerve block to be applied with ultrasound guidance.
  Interventions: Other: Interscalene block
- suprascapular and infraclavicular nerve block (Active Comparator): preoperative suprascapular and infraclavicular nerve block to be with ultrasound guidance
  Interventions: Other: suprascapular and infraclavicular nerve block

INTERVENTIONS:
Other: Interscalene block — 30 minutes before anaesthesia induction interscalene nerve block will be applied with ultrasound guidance with %0,25 bupivacain 20 cc .The sham block consisted of after patients were placed in the lateral decubitus position skin preparation, ultrasound scanning of the suprascapular region, and a dry-needling, all performed to preserve patient blinding in the ISB group patients.
  Arms: Interscalene nerve block
Other: suprascapular and infraclavicular nerve block — 30 minutes before anaesthesia induction suprascapular with %0,25 bupivacain 10 cc .and infraclavicular nerve block with %0,25 bupivacain 10 cc will be applied with ultrasound guidance
  Arms: suprascapular and infraclavicular nerve block

SUMMARY:
It is compared that combined suprascapular and infraclavicular nerve blocks to interscalene nerve block for clinical outcomes after shoulder surgery

DETAILED DESCRIPTION:
In this study, the investigators planned to investigate postoperative pain, analgesic dosage, respiratory effects of the block and side effects of patients undergoing general anaesthesia after arthroscopic shoulder surgery under preoperative interscalene nerve block or suprascapular + infraclavicular nerve block.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for elective shoulder surgery under general anesthesia with suprascapular + infraclavicular nerve block or interscalene nerve block for any reason ASA 1-3 patients

Exclusion Criteria:

* Diabetes
* coagulopathy
* local anesthetic allergy
* chronic opioid users
* neurological deficit of the surgical limb
* obstructive or restrictive pulmoner disease
* inability to understand pain scores

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2019-09-30 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
postoperative pain: numeric rating scale (NRS) | postoperative 30. minute, 4. hour, 8.hour,12. hour, 24. hour, 48. hour
  postoperative pain will be evaluated by numeric rating scale (NRS) .

SECONDARY OUTCOMES:
phrenic nerve paralysis evaluated with ultrasound | thirty minutes after the nerve block
  Thirty minutes after the block, M-mode ultrasound examination of the ipsilateral hemidiaphragm was performed to measure diaphragmatic excursion.

CONTACTS AND LOCATIONS:
Locations (1):
- Diskapi Yildiim Beyazit Eduation and Research Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No